CLINICAL TRIAL: NCT00993174
Title: Amount of Surgery for Esotropia Under Topical Anesthesia
Brief Title: Surgery for Esotropia Under Topical Anesthesia
Acronym: SETTA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitario Ramon y Cajal (Other)
Collaborators: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Jaime Tejedor, Hospital Ramón y Cajal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SETTA
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2010-05

CONDITIONS: Esotropia
MeSH Terms: conditions — Esotropia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topical anesthesia (Experimental): Patients undergo strabismus surgery for esotropia using topical anesthesia (instillation of drops plus gel)
  Interventions: Procedure: Topical strabismus surgery
- Sub-Tenon's anesthesia (Active Comparator): Patients undergo surgery for strabismus (esotropia) using sub-Tenon's administration of anesthetic (xylocaine)
  Interventions: Procedure: Sub-Tenon's strabismus surgery

INTERVENTIONS:
Procedure: Topical strabismus surgery — Surgery is carried out after instilling drops for anesthesia and administering lidocaine gel during the procedure
  Arms: Topical anesthesia
Procedure: Sub-Tenon's strabismus surgery — Surgery is carried out after sub-Tenon's injection of xylocaine
  Arms: Sub-Tenon's anesthesia

SUMMARY:
Adult patients requiring surgery for esotropia will be randomized to surgery under topical anesthesia or sub-Tenon's anesthesia. Amount of surgery required with the two anesthetic procedures will be compared. Motor and sensory outcome of the two treatment groups will also be compared.

ELIGIBILITY:
Inclusion Criteria:

* Esotropia deviation angle equal to or lower than 45 prism dioptres (requiring one or two-muscle surgery)
* Visual acuity at least 20/40 in each eye
* Cooperation for topical anesthesia

Exclusion Criteria:

* Paretic or restrictive strabismus
* Previous eye muscle surgery
* Significant eye disease other than strabismus

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2004-05; Primary Completion 2009-06 (Actual); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Amount of surgery required in mm and mm/degree of deviation angle | Immediate

SECONDARY OUTCOMES:
Motor (deviation angle) and stereoacuity outcome | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Tejedor, MD, PhD, Principal Investigator — Hospital Universitario Ramon y Cajal
Locations (1):
- Hospital Univ Ramón y Cajal, Madrid, Madrid, Spain